CLINICAL TRIAL: NCT04952649
Title: The Ability of Peripheral Perfusion Index To Detect Changes of Hemodynamics in Patients With Pacemaker：a Prospective Study
Brief Title: The Ability of Peripheral Perfusion Index To Detect Changes of Hemodynamics in Patients With Pacemaker
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PITCH
Record Dates: First submitted 2021-06-18; First posted 2021-07-07 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Pacemaker Dependence
Keywords: peripheral perfusion index; cardiac output; stroke volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pacemaker dependent patients after cardiac surgery: Pacemakers are widely used in cardiotomy patients, while it's common that the patients happen to be pacemaker dependent. When the doctor decides to set the heart rate of the pacemaker, we record the hemodynamic parameters and peripheral perfusion index from 70-80-90-100-110 bpm.

SUMMARY:
Pacemakers are widely used in postcardiotomy patients to avoid severe arrhythmia. The peripheral perfusion index (PI) has been considered as an effective parameter evaluating the circulation. In this study, investigators aim to avaluate the ability of peripheral perfusion index to detect changes of hemodynamics in postcardiotomy patients with pacemakers.

DETAILED DESCRIPTION:
Pacemakers are widely used in postcardiotomy patients to avoid severe arrhythmia. The peripheral perfusion index (PI) has been considered as an effective parameter evaluating the circulation. In this study, investigators aim to evaluate the ability of peripheral perfusion index to detect changes of hemodynamics (cardiac output or storke volume,et al) in postcardiotomy patients with pacemakers.

ELIGIBILITY:
Inclusion Criteria:

* age >=18 years old;
* postcardiotomy
* placement of temportary pacemaker during the surgery
* dependence of pacemaker (abscence of autonomic cardiac rhythm）

Exclusion Criteria:

* hemodynamic unstable （high dose of vasoactive drugs）
* fingers ischemia, cannot monitor the peripheral perfusion index

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pacemakers are widely used in post-cardiotomy patients, while it's common that some patients may be pacemaker dependent. We choose these patients who has been placed with temportary pacemaker during the cardic surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | During the study procedure
  Measurement of cardiac output by Flotrac ,the metric is L/min.
stroke volume | During the study procedure
  Measurement of stroke volume by Flotrac ,the metric is ml.
Peripheral perfusion index | During the study procedure
  Measurement of Peripheral perfusion index by masimo radical.

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, MD PhD, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Background] Bazaraa H, Roby S, Salah E, Algebaly H. Assessment of Tissue Perfusion Using the Peripheral Perfusion Index and Lactate Clearance in Shock in Pediatric Patients. Shock. 2021 Dec 1;56(6):933-938. doi: 10.1097/SHK.0000000000001811. PMID 34014888
- [Background] Abdel-Ghaffar HS, Abdel-Wahab AH, Roushdy MM. Using the Perfusion Index to predict changes in the depth of anesthesia in children compared with the A-line Autoregression Index: an observational study. Braz J Anesthesiol. 2024 Sep-Oct;74(5):744169. doi: 10.1016/j.bjane.2021.04.030. Epub 2021 May 12. PMID 33991553